CLINICAL TRIAL: NCT07365774
Title: The Role of the "Let's Go to the Dentist!" Video Modelling and Dental Determinants on Dental Anxiety in Children
Brief Title: Video Modelling and Dental Determinants on Dental Anxiety in Children
Acronym: VMDDAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wisnu Fadila (Other)
Collaborators: Badan Riset dan Inovasi Nasional BRIN, Indonesia (Unknown)
Responsible Party: Sponsor-Investigator, Wisnu Fadila, Doctoral Candidate, Universitas Padjadjaran
Organization: Universitas Padjadjaran (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DENT-202601.01
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dental Anxiety
Keywords: Dental Anxiety; Video Modelling; Children; Caries Experience; Dental Visits; Oral Health Knowledge; Sociodemographic Factors; Modified Dental Anxiety Scale

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Modelling (Experimental): Children complete baseline Modified Dental Anxiety Scale Integrated with Facial Image Scale assessment (MDAS+FIS). They then view the "Let's Go to the Dentist!" video (2 minutes 37 seconds). MDAS+FIS is assessed immediately afterward (posttest 1). After a 30-minute wait period, children view the same video again. MDAS+FIS is assessed immediately afterward (posttest 2).
  Interventions: Behavioral: "Let's Go to the Dentist!" Video Modelling
- Educational Video (Placebo Comparator): Children complete baseline Modified Dental Anxiety Scale Integrated with Facial Image Scale (MDAS+FIS) assessment. They then view the "Let's Brush Our Teeth!" video (2 minutes 16 seconds). MDAS+FIS is assessed immediately afterward (posttest 1). After a 30-minute wait period, children view the same video again. MDAS+FIS is assessed immediately afterward (posttest 2).
  Interventions: Behavioral: "Let's Brush Our Teeth!" General Dental Education Video
- Control (No Intervention): Children complete baseline Modified Dental Anxiety Scale Integrated with Facial Image Scale (MDAS+FIS) assessment. They wait 30 minutes with no video intervention. MDAS+FIS is assessed at matching time points (posttest 1 equivalent and posttest 2 equivalent).

INTERVENTIONS:
Behavioral: "Let's Go to the Dentist!" Video Modelling — A 2 minutes 37 seconds video depicting a girl demonstrating calm and cooperative behaviour throughout a complete dental visit, from arrival through discharge. Content includes:
  * Greeting dental staff calmly
  * Sitting cooperatively in dental chair
  * Responding positively to instructions
  * Maintaining calm body language during examination
  * Completing all procedures without distress
  * Leaving with positive expressions
  Arms: Video Modelling
Behavioral: "Let's Brush Our Teeth!" General Dental Education Video — A 2 minutes 16 seconds educational video of a boy demonstrating correct toothbrushing technique and basic dental hygiene practices.
  Content includes:
  * Proper toothbrush selection
  * Correct toothbrushing method
  * Duration of brushing
  * Interdental cleaning
  * Fluoride use
  Arms: Educational Video

SUMMARY:
The goal of this clinical trial is to determine if video modelling reduces dental anxiety in children aged 8-12 years in Depok City. The main questions it aims to answer are: Does video modelling exposure significantly lower dental anxiety levels compared to educational video or control groups? Do family sociodemographic factors, dental health knowledge, dental visit patterns, and caries experience contribute to children's dental anxiety? Researchers compare anxiety scores of the video modelling group to the educational video group and control group (no intervention) to assess anxiety reduction effects before and after controlling for confounding factors. Children aged 8-12 years are the participants. Enumerators interview them using the Modified Dental Anxiety Scale Integrated with Facial Image Scale (MDAS+FIS) before and after each intervention, while children watch assigned videos: video modelling (twice), educational video (twice), or none (control). Enumerators record all responses. Children also undergo World Health Organization Decayed, Missing, and Filled Teeth (WHO DMFT/dmft) index dental exams plus interviews about dental knowledge, practices, caries complaints, and visit patterns. Parents complete separate interviews and surveys about family sociodemographics, their own dental knowledge and practice, and their children's dental knowledge, practices, visits, and caries experience.

DETAILED DESCRIPTION:
Dental problems affect children worldwide due to sociodemographic factors, high sugar intake, limited access, urbanization, and lifestyle changes, particularly in low and middle income countries. Indonesia's Riset Kesehatan Dasar/Basic Health Research (Riskesdas) 2018 documented 67.3% prevalence among children aged 5-9 years and 55.6% among 10-14 years with only 14.6% and 9.4% accessing professional care respectively, highlighting dental anxiety as a key mediator alongside established risk factors. Family and school environments critically shape children's dental health attitudes, supporting early promotive preventive interventions.

This study tests video modeling, a safe, scalable nonpharmacologic approach leveraging observational learning, against placebo and control conditions. The experimental intervention demonstrates sequential prosocial behaviors through a child model, including calm greeting of dental staff, positive responses to instructions, procedural tolerance without distress, and satisfied departure.

The design evaluates repeated exposure effects, specifically two viewings with 30 minute interval, within urban Depok elementary schools representing diverse socioeconomic contexts. Parental interviews provide additional perspectives alongside quantitative outcomes on dental health determinants, informing national policy translation

ELIGIBILITY:
Inclusion Criteria:

1. Schoolchildren aged 8-12 years old at time of enrolment
2. Resident of Depok City, West Java, Indonesia
3. Currently enrolled in participating elementary school
4. Parent/legal guardian able to provide written informed consent
5. Child able to provide verbal assent to participate
6. Willing and able to complete study assessments

Exclusion Criteria:

1. Currently receiving orthodontic treatment
2. Reside outside Depok City boundaries (verified post-assessment)
3. Age criteria violation (outside 8-12 year range at assessment)
4. Parent/caregiver unavailable for parent questionnaire interview
5. Incomplete child questionnaire responses on outcome measures
6. Institutional residence (orphanage, boarding school)
7. Inability to provide informed consent/assent

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 496 (Actual)
Dates: Start 2024-10-26 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dental Anxiety Level | Baseline to post-intervention 1 (immediately after first video exposure), then to post-intervention 2 (immediately after second video exposure, 30 minutes after first post-assessment).
  Change in dental anxiety scores assessed by the Modified Dental Anxiety Scale Integrated with Facial Image Scale (MDAS+FIS). The MDAS+FIS consists of 5 items scored from 1 to 5, giving a total score range of 5 (lowest anxiety) to 25 (highest anxiety), and higher scores indicate worse (greater) dental anxiety levels.
Dental Health Determinants Assessment | Baseline
  Structured assessment of:
  * Sociodemographic factors (age, sex, grade, birth order, parental education, family income, school type)
  * Dental visit patterns (frequency past 12 months)
  * Dental health knowledge (toothbrushing frequency, time, caries cause)
  * Caries experience using World Health Organization Decayed, Missing, and Filled Teeth (WHO DMFT/dmft) index per WHO Oral Health Surveys Basic Methods, 2013.

CONTACTS AND LOCATIONS:
Overall Officials: Wisnu Fadila, DDS, MSR, Principal Investigator — Universitas Padjadjaran
Locations (6):
- Indonesia (6):
  - Sekolah Dasar Ar-Rahman Islamic School (Ar-Rahman Islamic Elementary School), Depok, West Java
  - Sekolah Dasar Islam Plus Darul Ulum (Darul Ulum Islamic Plus Elementary School), Depok, West Java
  - Sekolah Dasar Negeri Cinere 1 (Cinere 1 Public Elementary School), Depok, West Java
  - Sekolah Dasar Negeri Gandul 1 (Gandul 1 Public Elementary School), Depok, West Java
  - Sekolah Dasar Negeri Krukut 1 (Krukut 1 Public Elementary School), Depok, West Java
  - Sekolah Dasar Negeri Pangkalan Jati 1 (Pangkalan Jati 1 Public Elementary School), Depok, West Java

IPD SHARING:
Plan to Share IPD: No
Prohibited by Indonesian law under Personal Data Protection Act 2022.